CLINICAL TRIAL: NCT06882252
Title: Increasing Lean Protein Intake in Preschool-age Children
Brief Title: Increasing Lean Protein Intake in Preschool-age Children and Assessing Effects on Cognition and Select Health Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sibylle Kranz, PhD, RDN (Other)
Responsible Party: Sponsor-Investigator, Sibylle Kranz, PhD, RDN, Associate Professor, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HSR231601
Record Dates: First submitted 2025-02-20; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Diet Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Diet modification: Low glycemic index diet Meal and snack are made with lean pork to reduce glycemic index of food consumed.
  Interventions: Other: Low glycemic index diet
- Control (No Intervention): Typically consumed meal and snack; high glycemic index

INTERVENTIONS:
Other: Low glycemic index diet — Replacement of typical meal/snack with lean pork containing meal/snack
  Arms: Intervention

SUMMARY:
The proposed project addresses the goal of exploring preschooler's ability to recognize changes in feelings of hunger/satiety based on consuming a snack and a meal (lunch/dinner) that are either based on the usual childcare center fare (control) or are based on lean meats (intervention), which will have a lower glycemic index.

ELIGIBILITY:
Inclusion Criteria:

* child 2-5 years old

Parent participants:

* Parents of at least one child aged 2-5 years old
* Parents can communicate in English.
* Parents in households who do not have a cultural/ religious reason to abstain from to consuming pork

Exclusion Criteria:

* Child participants:
* Food allergies
* Taking medication that affects food intake (such as stimulant medications),
* Children with diabetes or impaired glucose control.
* Children with digestive disease (such as Crohn's)
* Dietary/religious preferences that exclude consumption of pork

Parent participants:

- Dietary/religious preferences that exclude consumption of pork

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic load of diet | 6 study days
  Estimated intake of glycemic load of meals and snacks consumed. Plate-waste method will be used to calculate total energy, GI, GL consumed at each meal and snack using disaggregated intake (in grams) and analysis using Nutrient Data System for Research (NDS-R) software.
Hunger/Satiety self-reported on 4-point scale | 6 study days
  Self-reported feelings of hunger or fullness using: 1 = Very hungry, 2 = A little hungry, 3 = A little full, 4 = Very full

SECONDARY OUTCOMES:
Blood pressure | 60 minutes after the meal.
  Measured blood pressure 60 minutes after the meal.
Blood glucose | 6 study days
  Blood glucose concentration 60 minutes after the meal. Measured using finger-stick and glucometer reading.
Executive function: focus and short-term memory | 6 study days
  Using the "track-it" game, children respond to visual cues.
Executive function: memory and focus | 6 study days
  Using KRISP, children respond to visual cues to assess focus and short-term memory
Executive Function: Focus and Concentration | 6 study days
  Using the "peg it" game, children are asked to use a small wooden hammer to tab the table surface. First, they repeat how many tabs the researcher demonstrated (1 or 2), then they are asked to tab the opposite, so if the researcher tabs once, they tab twice and when the researcher tabs twice, they tab once.
Executive Function: Concentration | 6 study days
  Using the happy-sad game, children sort small playing cards with happy or sad faces on them to align with the verbal cue of the researcher, or to put down the opposite card.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot and feasibility study and subjects may be identified if individual participant data is shared.

REFERENCES:
- [Background] Varley BJ, Nasir RF, Skilton MR, Craig ME, Gow ML. Early Life Determinants of Vascular Structure in Fetuses, Infants, Children, and Adolescents: A Systematic Review and Meta-Analysis. J Pediatr. 2023 Jan;252:101-110.e9. doi: 10.1016/j.jpeds.2022.08.033. Epub 2022 Aug 24. PMID 36029824
- [Background] Mikkila V, Rasanen L, Raitakari OT, Pietinen P, Viikari J. Consistent dietary patterns identified from childhood to adulthood: the cardiovascular risk in Young Finns Study. Br J Nutr. 2005 Jun;93(6):923-31. doi: 10.1079/bjn20051418. PMID 16022763